CLINICAL TRIAL: NCT00739466
Title: Intravenous Liposomal Alendronate Infusion in Subjects Undergoing Bare Metal Coronary Stent Implantation
Brief Title: Biorest Liposomal Alendronate With Stenting sTudy (BLAST)
Acronym: BLAST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BIOrest Ltd. (Industry)
Collaborators: Baim Institute for Clinical Research (Other); Cardiovascular Research Foundation, New York (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LA-II-01
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Coronary Artery Stenosis
Keywords: Liposomal Alendronate; Percutaneous coronary intervention; Coronary stenting; de novo stenotic lesions; Native coronary arteries; Restenosis; Bare metal stent; Presillion CoCr coronary stent
MeSH Terms: conditions — Coronary Stenosis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- low dose (Experimental): Liposomal Alendronate dose of 0.001 mg
  Interventions: Drug: Liposomal Alendronate
- high dose (Experimental): Liposomal Alendronate dose of 0.01 mg
  Interventions: Drug: Liposomal Alendronate
- placebo (Placebo Comparator): IV saline infusion
  Interventions: Drug: Saline infusion (placebo)

INTERVENTIONS:
Drug: Liposomal Alendronate — IV in a single low dose during the index procedure (coronary stent implantation) over 2 hours
  Other Names: LA
  Arms: low dose
Drug: Liposomal Alendronate — IV in a single high dose during the index procedure (coronary stent implantation) over 2 hours
  Other Names: LA
  Arms: high dose
Drug: Saline infusion (placebo) — IV saline infusion during the index procedure (coronary stent implantation) over 2 hours
  Other Names: Saline
  Arms: placebo

SUMMARY:
The main objective of this study is to assess the safety and efficacy of Liposomal Alendronate in the treatment of de novo stenotic lesions in native coronary arteries in a population undergoing PCI with implantation of a bare metal stent.

Study hypothesis: Liposomal Alendronate will reduce in-stent restenosis as compared to placebo.

DETAILED DESCRIPTION:
This is a Phase II dose-finding, randomized, multi-center, prospective, double blind clinical study. Subjects undergoing percutaneous coronary intervention (PCI) with the Presillion™ CoCr bare metal stent will be randomized into three groups and administered (in a single dose intravenously (IV) through a peripheral venous catheter) either: low dose Liposomal Alendronate of 0.001 mg, high dose Liposomal Alendronate of 0.01 mg, or placebo (IV saline infusion) on a 1:1:1 basis.

All subjects will undergo angiographic follow-up at 6 months and 110 subjects enrolled from pre-specified sites will undergo intravascular ultrasound (IVUS) at baseline and follow-up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is eligible for percutaneous coronary intervention .
2. Subject is an acceptable candidate for coronary artery bypass graft surgery.
3. Subject has stable angina pectoris
4. Subject is a candidate for elective stenting of up to 2 lesions.

Exclusion Criteria:

General

1. Any planned elective surgery or percutaneous intervention within 6 months post-procedure.
2. A previous coronary interventional procedure of any kind within 30 days prior to the procedure.
3. Subject requires a staged procedure of either the target or any non-target vessel within 9 months post-procedure.
4. Any drug eluting stent (DES) deployment within the past 12 months.
5. Any planned drug eluting stent (DES) deployment during the procedure associated with this study or within 3 months following the index procedure.
6. Known hypersensitivity or contraindication to aspirin or clopidogrel or a sensitivity to contrast media, which cannot be adequately pre-medicated
7. Concurrent medical condition with a life expectancy of less than 12 months.
8. Documented left ventricular ejection fraction (LVEF) < 25% at the most recent evaluation.
9. Evidence of ST elevated myocardial infarction (STEMI) or non-STEMI with troponin (cTn) levels greater than or equal to 3 times the normal limit at any time within 72 hours of the intended trial procedure.
10. History of cerebrovascular accident or transient ischemic attack in the last 6 months.
11. Leukopenia .
12. Neutropenia
13. Thrombocytopenia
14. Serum creatinine level >2.5 mg/dl within 7 days prior to index procedure.
15. History of bleeding diathesis or coagulopathy or inability to accept blood transfusions.
16. Known hypersensitivity or contraindication to aspirin, heparin or bivalirudin, clopidogrel and ticlopidine, cobalt, nickel, L-605 Cobalt chromium alloy, Alendronate or sensitivity to contrast media, which cannot be adequately pre-medicated.
17. History of severe:Gastrointestinal disease,Immunodeficiency,Bone diseases

Angiographic Exclusion Criteria

1. Unprotected left main coronary artery disease (obstruction greater than 50% in the left main coronary artery that is not protected by at least one non-obstructed bypass graft to the LAD or Circumflex artery or a branch thereof).
2. Any previous stent placement within 15 mm (proximal or distal) of the target lesion(s).
3. Target vessel exhibiting lesions with greater than 60% diameter stenosis outside of a range of 5 mm proximal and distal to the target lesion(s) based on visual estimate or on-line QCA.
4. Target lesion(s) exhibiting an intraluminal thrombus (occupying >50% of the true lumen diameter) at any time.
5. Lesion location that is aorto-ostial or within 5 mm of the origin of the left anterior descending (LAD) or left circumflex (LCX).
6. The target lesion(s) requires treatment with a device other than PTCA prior to stent placement (such as, but not limited to, directional coronary atherectomy, excimer laser, rotational atherectomy, etc.).
7. Target lesion(s) with side branches > 2.0mm in diameter.
8. Target lesion(s) involving a bifurcation (either stenosis of both main vessel and major branch or stenosis of just major branch).
9. Target lesion(s) with severe calcification.
10. Target vessel exhibiting excessive tortuosity that may impede stent delivery and deployment at target lesion(s).
11. Target lesion(s) located in a native vessel distal to an anastomosis with a saphenous vein graft or a left/right internal mammary artery (LIMA/RIMA) bypass.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2008-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
In-stent late loss: measured at 6 months post-procedure as determined by quantitative coronary angiography (QCA). | 6 months post-procedure

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | at 30, 180 and 360 days as well as yearly through 5 years post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Prof Shmuel Banai, MD, Principal Investigator — The Tel Aviv Sourasky Medical Center
Locations (12):
- Israel (12):
  - Hillel Yaffe Medical Center, Hadera
  - Bnei Zion Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Western Galilee Hospital, Nahariya, Nahariya
  - Rabin Medical Center, Petah Tikva
  - The Baruch Padeh Medical Center, Poriya, Poria – Neve Oved
  - Sheba Medical Center, Tel Hashomer, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - The Tel Aviv Sourasky Medical Center, Tel Aviv

REFERENCES:
- [Derived] Banai S, Finkelstein A, Almagor Y, Assali A, Hasin Y, Rosenschein U, Apruzzese P, Lansky AJ, Kume T, Edelman ER. Targeted anti-inflammatory systemic therapy for restenosis: the Biorest Liposomal Alendronate with Stenting sTudy (BLAST)-a double blind, randomized clinical trial. Am Heart J. 2013 Feb;165(2):234-40.e1. doi: 10.1016/j.ahj.2012.10.023. Epub 2012 Dec 11. PMID 23351827